CLINICAL TRIAL: NCT00241332
Title: Prophylaxis Against Postoperative Pain After Orthopedic Surgery: Does it Help to Give Fentanyl Before Start of Remifentanil/Propofol Based Anesthesia?
Brief Title: Postoperative Pain After Orthopedic Surgery: Does it Help to Give Fentanyl Before Start of Remifentanil Based Anesthesia?
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Ullevaal University Hospital (Other)
Collaborators: University of Oslo (Other)
Organization: Oslo University Hospital (Other)
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: 510-05165
Record Dates: First submitted 2005-10-17; First posted 2005-10-18 (Estimated); Last update posted 2011-07-06 (Estimated); Status verified 2005-09

CONDITIONS: Pain, Postoperative
Keywords: pain; hyperalgesia; drug tolerance; remifentanil; fentanyl; Anterior Cruciate Ligament; Posterior Cruciate Ligament; Medial Collateral Ligament, Knee
MeSH Terms: conditions — Pain, Postoperative; Pain; Hyperalgesia | interventions — Fentanyl

INTERVENTIONS:
Drug: fentanyl

SUMMARY:
The aim of this trial is to examine the possibility that fentanyl 1,5 µgr/kg given intravenously (i.v.) before the start of remifentanil infusion for anesthesia gives less development of tolerance/hyperalgesia postoperative than fentanyl given at the end of surgery (the traditional method).

DETAILED DESCRIPTION:
Postoperative pain can contribute to reduction in the patient's well-being and, if it is pronounced, delayed rehabilitation and an increase in the total cost for nursing and treatment.

Experimental studies has shown that infusion of remifentanil over some period of time, can result in acute opioid tolerance and hyperalgesia (1-2).

One clinical trial has shown that intraoperative infusion of remifentanil gives acute opioid tolerance with subsequent increased postoperative pain and increased opioid consume postoperative (3).

The development of opioid tolerance probably has several mechanisms. One topical mechanism is opioid induced influence of N-methyl-d-aspartate (NMDA)-receptor and its intracellular second-messenger-systems. This results in central sensitization to pain stimulus in the dorsal horn and the brain (4-5), with following development of hyperalgesia.

Several strategies can be successful to reduce or prevent opioid induced hyperalgesia, for example NMDA-receptor antagonists, alfa-2 agonists, opioid rotation or combination of opioids with different receptor selectivity (6-8).

The theoretical background for pre-treating the opioid receptor with an other opioid (fentanyl) that gives less tendency to hyperalgesia than remifentanil, is that it can reduce the development of tolerance and hyperalgesia of remifentanil.

The aim of this trial is to examine the possibility that i.v. administration of fentanyl 1,5 µgr/kg before start of remifentanil infusion for anesthesia gives less development of tolerance/hyperalgesia postoperative than fentanyl given in the end of surgery (the traditional method).

This is to be measured by less pain postoperative (VAS, visual analog scale, and a five point verbal rating scale) and less fentanyl consumed (measured by using PCA).

Literature:

1. Vinik HR, Kissin I (1998) Rapid development of tolerance to analgesia during remifentanil infusion in human. Anesth Analg 86:1307-1311.
2. Angst MS, Koppert W, Pahl I, Clark JD, Schmelz M (2003) Short-term infusion of the µ-opioid agonist remifentanil in humans causes hyperalgesia during withdrawal. Pain 106:49-57.
3. Guignard et al. (2000) Acute opioid tolerance: intraoperative remifentanil increases postoperative pain and morphine requirement. Anesthesiology 93:409-417.
4. Larcher A, Laulin JP, Celerier E, Le Moal M, Simonnet G (1998) Acute tolerance associated with a single opioid administration: involvement of N-methyl-D-aspartate-dependent pain facilitatory systems. Neuroscience Vol 84:583-589.
5. Celerier E, Laulin J, Larcher A, Le Moal M, Simonnet G (1999) Evidence for opiate-activated NMDA processes masking opiate analgesia in rats. Brain Research 849:18-25.
6. Celerier E, Rivat C, Jun Y, Laulin JP, Larcher A, Reynier P, Simonnet G(2000) Long-lasting hyperalgesia induced by fentanyl in rats: preventive Effect of ketamin. Anesthesiology 92:465-472.
7. Bie B, Fields HL, Williams JT, Pan ZZ (2003) Roles of a alfa-1 and alfa-2-adrenoreceptors in the nucleus raphe magnus in opioid analgesia and opioid abstinence-induced hyperalgesia. Journal of Neuroscience 23:7950-7957.
8. Mao J, Prince DD, Caruso F, Mayer DJ (1996) Oral administration of dextromethorphan prevents the development of morphine tolerance and dependence in rats. Pain 67:361-368.

ELIGIBILITY:
Inclusion Criteria:

* Women and men > 18 years.
* Informed consent.
* Elective day-orthopedic surgery: damage to anterior cruciate ligament and/or posterior cruciate ligament with or without medial collateral ligament.

Exclusion Criteria:

* Patients who use nonsteroidal anti-inflammatory drugs (NSAID's) or are allergic to NSAID's.
* Patients using steroids, anti-emetics, drugs or opioids.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100
Dates: Start 2005-10; Study Completion 2006-07 (Actual)

PRIMARY OUTCOMES:
Less use of postoperative opioids
Less visual analog scale (VAS) and verbal rating scale (VRS) in the treatment group

CONTACTS AND LOCATIONS:
Overall Officials: Johan Ræder, Prof.MD,Phd, Study Director — Ullevaal University Hospital
Locations (1):
- Ullevaal University Hospital, Oslo, Oslo County, Norway